CLINICAL TRIAL: NCT06702644
Title: Safety and Efficacy of Remote Ischemic Conditioning in Patients with Chronic Internal Carotid Artery Occlusion Receiving Hybird Surgery: a Pilot, Randomized Controlled Trial
Acronym: SERIC-HS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Vice president of The First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SERIC-HS
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Carotid Artery Occlusion
Keywords: RIC; remote ischemic conditioning; carotid artery occlusion; hybird surgery; interventional surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RIC (Active Comparator): Remote ischemic conditioning (RIC) is induced by 5 cycles of 5 min of bilateral upper limbs ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mmHg. RIC will be conducted twice daily for 6 consecutive days after enrollment.
  Interventions: Device: Remote ischemic conditioning
- Sham RIC (Placebo Comparator): Sham remote ischemic conditioning (RIC) is induced by 5 cycles of 5 min of bilateral upper limbs ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mmHg. Sham RIC will be conducted twice daily for 6 consecutive days after enrollment.
  Interventions: Device: Sham remote ischemic conditioning

INTERVENTIONS:
Device: Remote ischemic conditioning — Remote ischemic conditioning: Remote ischemic conditioning (RIC) is induced by 5 cycles of 5 min of bilateral upper limbs ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 200 mmHg.
  Arms: RIC
Device: Sham remote ischemic conditioning — Sham remote ischemic conditioning (RIC) is induced by 5 cycles of 5 min of bilateral upper limbs ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 60 mmHg.
  Arms: Sham RIC

SUMMARY:
The purpose of this study is to explore the safety and efficacy of remote ischemic conditioning in patients with internal carotid artery occlusion receiving hybird surgery.

DETAILED DESCRIPTION:
In this study, 60 patients with internal carotid artery occlusion receiving hybird surgery are included in our center in China. The experimental group will receive basic treatment and remote ischemic conditioning for 200mmHg, 2 times per day for 6 consecutive days. The control group will receive basic treatment and remote ischemic conditioning control for 60mmHg, 2 times per day for 6 consecutive days. Two groups will be followed up for 90 days to evaluate the safety and efficacy of remote ischemic conditioning in patients with internal carotid artery occlusion receiving hybird surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years, regardless of sex
* Patients with chronic carotid artery occlusion who are going to undergo hybird surgery
* Can cooperate with and complete brain magnetic resonance imaging (MRI) examination
* Signed and dated informed consent is obtained

Exclusion Criteria:

* Hemorrhagic stroke
* Severe cardiac dysfunction or arrhythmia
* Uncontrolled hypertension (defined as systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg, despite medication taken at enrollment)
* Severe hepatic and renal dysfunction (defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥3 times higher than the upper limit of the normal range, creatinine >265umol/l (3mg/dl))
* The patients who have the contraindication of remote ischemic conditioning treatment, such as severe soft tissue injury, fracture or vascular injury in the upper limb. Acute or subacute venous thrombosis, arterial occlusive disease, subclavian steal syndrome, etc.
* Pregnant or lactating women
* He/She is participating in other clinical research or has participated in other clinical research or has participated in this study within 3 months prior to admission
* Other conditions that the researchers think are not suitable for the group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with new Diffusion Weighted Imaging (DWI) - positive lesions on post-treatment magnetic resonance imaging (MRI) Scans. | 6 days
  Patients will undergo magnetic resonance imaging (including DWI) at baseline and 6 days after randomization.

SECONDARY OUTCOMES:
The number of new Diffusion Weighted Imaging (DWI)-positive lesions on post-treatment magnetic resonance imaging (MRI) Scans. | 6 days
  Patients will undergo magnetic resonance imaging (including DWI)at baseline and 6 days after randomization.
The volume of new Diffusion Weighted Imaging (DWI)-positive lesions on post-treatment magnetic resonance imaging (MRI) Scans. | 6 days
  Patients will undergo magnetic resonance imaging(including DWI) at baseline and 6 days after randomization.
Number of patients with cerebrovascular events, cardiovascular events or death | 90±7 days
  Cerebrovascular events include ischemic stroke, transient ischemic attack (TIA), cerebral hemorrhage. Cardiovascular events include angina and myocardial infarction. Death include all-cause of death.
Proportion of patients with any side effects of RIC treatment. | 6 days
  The side effects referred to any side effects of RIC or sham RIC treatment, not including the sides effect of medications or hybrid surgery.
Proportion of patients with any adverse events（including serious adverse events) | 90±7 days
  Adverse events due to any cause after enrollment of subjects in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yang, MD, PhD, Study Chair — Neuroscience Center, Department of Neurology, The First Hospital of Jilin University

IPD SHARING:
Plan to Share IPD: No